CLINICAL TRIAL: NCT03933332
Title: Correlation Between Muscle Thickness and Inflammation With Ventilator Length of Use in Critically Ill Patients: Study on Diaphragm Thickness, Rectus Femoris and Biceps Brachii Cross-sectional Area, and C-reactive Protein Level
Brief Title: Correlation Between Muscle Thickness and Inflammation With Ventilator Use in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, MD, PhD, Anesthesiologist Consultant, Indonesia University
Other Study IDs: IndonesiaUAnes036
Record Dates: First submitted 2019-04-27; First posted 2019-05-01 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Ventilation Therapy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ventilator length of use: measured in days
  Interventions: Other: Diaphragm thickness; Other: Cross-sectional area of rectus femoris muscle; Other: Cross-sectional area of biceps brachii; Diagnostic Test: C-Reactive Protein (CRP) Level

INTERVENTIONS:
Other: Diaphragm thickness — measured at apposition zone using ultrasonography in mm
Other: Cross-sectional area of rectus femoris muscle — measured at lower one-third line between Spina iliaca anterior inferior (SIAI) and upper border femur patella using ultrasonography in cm^2
Other: Cross-sectional area of biceps brachii — measured at biceps brachii muscle using ultrasonography in cm^2
Diagnostic Test: C-Reactive Protein (CRP) Level — quantitative CRP using ELISA method in mcg/mL

SUMMARY:
Decrease thickness of diaphragm muscle, cross-sectional area of rectus femoris and biceps brachii muscle, and increase in CRP would affect ventilator length of use in critically ill patients in ICU

ELIGIBILITY:
Inclusion Criteria:

* Patients who had Modified Rankin Score < 4 in 1 month before admitted into ICU

Exclusion Criteria:

* Pregnant women
* Patients who had intubation more than 24 hours before admitted at ICU Cipto Mangunkusumo Hospital
* Patients who had a history or prior to thoracic or heart surgery 14 days before admission
* Patients who had severe peripheral muscle dysfunction
* Patients who had a history of admission in hospital for more than 2 weeks on the last 3 months
* Patients who predicted will be using ventilator for less than 4 days
* Patients who suffered acute respiratory distress syndrome (ARDS) with a ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) less than 200
* Patients who declined to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically-ill patients admitted to Intensive Care Units of Cipto Mangunkusumo Hospital using ventilator on October 2018 - December 2018
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in diaphragm thickness with ventilator length of use | 30 days from admission
  Correlation between changes in diaphragm thickness with ventilator length of use: < 7 days or >7 days
Correlation between changes in cross-sectional area of rectus femoris muscle with ventilator length of use | 30 days from admission
  Correlation between changes in cross-sectional area of rectus femoris muscle with ventilator length of use: < 7 days or >7 days
Correlation between changes in cross-sectional area of biceps brachii muscle with ventilator length of use | 30 days from admission
  Correlation between changes in cross-sectional area of biceps brachii muscle with ventilator length of use: < 7 days or >7 days
Correlation between changes in quantitative C-reactive protein (CRP) level with ventilator length of use | 30 days from admission
  Correlation between changes in quantitative C-reactive protein (CRP) level with ventilator length of use: < 7 days or >7 days

SECONDARY OUTCOMES:
Ventilator length of use | 30 days from admission
  duration of first ventilator use until patient is extubated or deceased: <7 days or >7 days
Changes in diaphragm thickness | 5 days from admission
  Measurement of diaphragm thickness from day 1 admission to ICU using ventilator to day 5 in mm
  Score for changes in diaphragm thickness:
  0 : no changes
  1. : decrease thickness of <20%
  2. : decrease thickness of >20%
Changes in cross-sectional area of rectus femoris muscle | 5 days from admission
  Measurement of cross-sectional area of rectus femoris muscle from day 1 admission to ICU using ventilator to day 5 in cm^2
  Score for changes in diaphragm thickness:
  0 : no changes
  1. : decrease cross-sectional area of <20%
  2. : decrease cross-sectional area of >20%
Changes in cross-sectional area of biceps brachii muscle | 5 days from admission
  Measurement of cross-sectional area of biceps brachii muscle from day 1 admission to ICU using ventilator to day 5 in cm^2
  Score for changes in diaphragm thickness:
  0 : no changes
  1. : decrease cross-sectional area of <20%
  2. : decrease cross-sectional area of >20%
Changes in quantitative C-reactive protein (CRP) levels | 5 days from admission
  Measurement of quantitative CRP from day 1 admission to ICU using ventilator to day 5 in mcg/mL
  Score for changes in diaphragm thickness:
  0 : no changes
  1. : increase in quantitative CRP <50%
  2. : increase in quantitative CRP >50%

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Mehta AB, Syeda SN, Wiener RS, Walkey AJ. Epidemiological trends in invasive mechanical ventilation in the United States: A population-based study. J Crit Care. 2015 Dec;30(6):1217-21. doi: 10.1016/j.jcrc.2015.07.007. Epub 2015 Jul 16. PMID 26271686
- [Background] Funk GC, Anders S, Breyer MK, Burghuber OC, Edelmann G, Heindl W, Hinterholzer G, Kohansal R, Schuster R, Schwarzmaier-D'Assie A, Valentin A, Hartl S. Incidence and outcome of weaning from mechanical ventilation according to new categories. Eur Respir J. 2010 Jan;35(1):88-94. doi: 10.1183/09031936.00056909. Epub 2009 Jun 18. PMID 19541716
- [Background] Hill AD, Fowler RA, Burns KE, Rose L, Pinto RL, Scales DC. Long-Term Outcomes and Health Care Utilization after Prolonged Mechanical Ventilation. Ann Am Thorac Soc. 2017 Mar;14(3):355-362. doi: 10.1513/AnnalsATS.201610-792OC. PMID 28033033
- [Background] Carson SS, Garrett J, Hanson LC, Lanier J, Govert J, Brake MC, Landucci DL, Cox CE, Carey TS. A prognostic model for one-year mortality in patients requiring prolonged mechanical ventilation. Crit Care Med. 2008 Jul;36(7):2061-9. doi: 10.1097/CCM.0b013e31817b8925. PMID 18552692
- [Background] Kim WY, Jo EJ, Eom JS, Mok J, Kim MH, Kim KU, Park HK, Lee MK, Lee K. Validation of the Prognosis for Prolonged Ventilation (ProVent) score in patients receiving 14days of mechanical ventilation. J Crit Care. 2018 Apr;44:249-254. doi: 10.1016/j.jcrc.2017.11.029. Epub 2017 Nov 23. PMID 29202432
- [Background] Clark PA, Inocencio RC, Lettieri CJ. I-TRACH: Validating A Tool for Predicting Prolonged Mechanical Ventilation. J Intensive Care Med. 2018 Oct;33(10):567-573. doi: 10.1177/0885066616679974. Epub 2016 Nov 30. PMID 27899470
- [Background] Clark PA, Lettieri CJ. Clinical model for predicting prolonged mechanical ventilation. J Crit Care. 2013 Oct;28(5):880.e1-7. doi: 10.1016/j.jcrc.2013.03.013. Epub 2013 May 14. PMID 23683556
- [Background] Latronico N, Gosselink R. A guided approach to diagnose severe muscle weakness in the intensive care unit. Rev Bras Ter Intensiva. 2015 Jul-Sep;27(3):199-201. doi: 10.5935/0103-507X.20150036. Epub 2015 Sep 15. No abstract available. PMID 26376161
- [Background] Latronico N, Piva S, McCredie V. Long-term implication of icu-acquired muscle weakness. In: Stevens RD, Hart N, Herridge MS, editors. Textbook of post-icu medicine. Oxford, UK: Oxford University Press; 2014. p. 259-68.
- [Background] Stevens RD, Marshall SA, Cornblath DR, Hoke A, Needham DM, de Jonghe B, Ali NA, Sharshar T. A framework for diagnosing and classifying intensive care unit-acquired weakness. Crit Care Med. 2009 Oct;37(10 Suppl):S299-308. doi: 10.1097/CCM.0b013e3181b6ef67. PMID 20046114
- [Background] Vincent JL, Norrenberg M. Intensive care unit-acquired weakness: framing the topic. Crit Care Med. 2009 Oct;37(10 Suppl):S296-8. doi: 10.1097/CCM.0b013e3181b6f1e1. PMID 20046113
- [Background] Hermans G, Van den Berghe G. Clinical review: intensive care unit acquired weakness. Crit Care. 2015 Aug 5;19(1):274. doi: 10.1186/s13054-015-0993-7. PMID 26242743
- [Background] Farhan H, Moreno-Duarte I, Latronico N, Zafonte R, Eikermann M. Acquired Muscle Weakness in the Surgical Intensive Care Unit: Nosology, Epidemiology, Diagnosis, and Prevention. Anesthesiology. 2016 Jan;124(1):207-34. doi: 10.1097/ALN.0000000000000874. PMID 26445385
- [Background] Latronico N, Herridge M, Hopkins RO, Angus D, Hart N, Hermans G, Iwashyna T, Arabi Y, Citerio G, Ely EW, Hall J, Mehta S, Puntillo K, Van den Hoeven J, Wunsch H, Cook D, Dos Santos C, Rubenfeld G, Vincent JL, Van den Berghe G, Azoulay E, Needham DM. The ICM research agenda on intensive care unit-acquired weakness. Intensive Care Med. 2017 Sep;43(9):1270-1281. doi: 10.1007/s00134-017-4757-5. Epub 2017 Mar 13. PMID 28289812
- [Background] Annetta MG, Pittiruti M, Silvestri D, Grieco DL, Maccaglia A, La Torre MF, Magarelli N, Mercurio G, Caricato A, Antonelli M. Ultrasound assessment of rectus femoris and anterior tibialis muscles in young trauma patients. Ann Intensive Care. 2017 Oct 6;7(1):104. doi: 10.1186/s13613-017-0326-x. PMID 28986861
- [Background] Nakanishi N, Oto J, Tsutsumi R, Iuchi M, Onodera M, Nishimura M. Upper and lower limb muscle atrophy in critically ill patients: an observational ultrasonography study. Intensive Care Med. 2018 Feb;44(2):263-264. doi: 10.1007/s00134-017-4975-x. Epub 2017 Nov 6. No abstract available. PMID 29110031
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Supinski GS, Morris PE, Dhar S, Callahan LA. Diaphragm Dysfunction in Critical Illness. Chest. 2018 Apr;153(4):1040-1051. doi: 10.1016/j.chest.2017.08.1157. Epub 2017 Sep 5. PMID 28887062
- [Background] Jorens PG, Schepens T. Ultrasound: a novel translational tool to study diaphragmatic dysfunction in critical illness. Ann Transl Med. 2016 Dec;4(24):515. doi: 10.21037/atm.2016.12.49. No abstract available. PMID 28149877